CLINICAL TRIAL: NCT05193552
Title: A Prospective Study of the Utility of Spirometry to Identify and Manage Immunoglobulin Replacement Dosage in Primary Antibody Deficiency in Patients with Potentially Reversible Airway Disease
Brief Title: Usage of Spirometry in Managing IgG Therapy in CVID with Airway Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Harry W. Schroeder, Jr., MD PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I300005696
Record Dates: First submitted 2021-08-06; First posted 2022-01-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Common Variable Immunodeficiency
MeSH Terms: conditions — Common Variable Immunodeficiency | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (No Intervention): 11 subjects will be treated for 6 months at their current dose of Hizentra
- Treatment Group (Experimental): 11 subjects will have their level of immunoglobulin replacement therapy increased by the equivalent of 0.05 gm/kg in dose per 4 weeks, adjusted for bioavailability as per manufacturer's instructions. On average, rounded up to the nearest gram, this will typically increase their dose of Hizentra by 2 gm per week.
  Interventions: Drug: Hizentra

INTERVENTIONS:
Drug: Hizentra — subjects level of immunoglobulin replacement therapy will be adjusted for bioavailability as per manufacturer's instructions
  Other Names: subcutaneous gammaglobulin therapy
  Arms: Treatment Group

SUMMARY:
Although there is evidence in the literature that gammaglobulin replacement therapy can lead to a reduction in the prevalence of pulmonary infection and improved lung function, there is no published study to guide immunologists regarding the use of spirometry in titrating IG therapy to assist in the management of immunodeficiency patients with regards to gammaglobulin replacement therapy.

The investigators propose to study the use of spirometry to identify patients that could potentially benefit from an increase in IGRT. The investigators will identify 22 common variable immune deficiency (CVID) study subjects on stable IGRT replacement therapy equivalent to 0.40 to 0.60 gm/kg per 4 weeks who have evidence of mild to moderate obstruction as assessed by an FEF25-75% between 50% and 80% of predicted. Patients who are on Hizentra will be preferentially recruited. Of these 22, 11 will be identified at random and treated for 6 months at their current dose (control population). The remaining 11 study subjects (treatment group) will have their level of IGRT increased by the equivalent of 0.05 gm/kg in dose per 4 weeks, adjusted for bioavailability as per manufacturer's instructions. On average, rounded up to the nearest gram, this will typically increase their dose of Hizentra by 2 gm per week.

DETAILED DESCRIPTION:
The key finding of the published retrospective study was that common variable immune deficiency (CVID) patients with moderate, presumed reversible, obstruction on stable, therapeutic doses of IgG who exhibited a decline in lung function from one clinic visit to the next responded to an increased dose of IgG with an improvement in lung function as assessed by spirometry.

The investigators now wish perform a clinical trial to assess whether primary antibody deficiency patients receiving IGRT who fit in this range of obstruction, i.e. an FEF25-75% that is 50-80% of predicted, will demonstrate an increase in lung function, as assessed by spirometry, after increasing the dose of IGRT. The presumption is that obstruction at this level is most likely due to the effects of subclinical infections that can be reduced or avoided by increasing the amount of gammaglobulin received by the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet criteria for common variable immune deficiency (CVID) who are on stable IGRT for at least 3 months and who have an FEF25-75% between 50% and 80% of predicted.
2. Patients who are already on Hizentra will be preferred.

Exclusion Criteria:

1. Age <21 or cannot perform spirometry.
2. Smokers with 20 pack years or more, and active smokers will not be included among the study subjects, but will be considered separately as an ancillary study.
3. Patients with specific antigen-specific antibody deficiencies or X-linked agammaglobulinemia on IGRT will not be included among the 20 study subjects, but will be considered separately in ancillary studies.
4. Patients with heart failure, TB, bronchiolitis, or lymphangioleiomyomatosis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
FEV1 at baseline | baseline
  Pulmonary function will be measured by forced expiratory volume in one second (FEV1) at baseline.
FEV1 at 3 months | 3 months
  Pulmonary function will be measured by forced expiratory volume in one second (FEV1) at three months into the study.
FEV1 at 6 months. | 6 months
  Pulmonary function will be measured by forced expiratory volume in one second (FEV1) at six months into the study.
FVC at baseline | baseline
  Pulmonary function will be measured by forced vital capacity (FVC) at baseline.
FVC at 3 months | 3 months
  Pulmonary function will be measured by forced vital capacity (FVC) at three months.
FVC at 6 months. | 6 months
  Pulmonary function will be measured by forced vital capacity (FVC) at six months.
FEF25-75% at baseline | baseline
  Pulmonary function will be measured by forced expiratory flow at 25 and 75% of the pulmonary volume (FEF25-75%) at baseline.
FEF25-75% at 3 months | 3 months
  Pulmonary function will be measured by forced expiratory flow at 25 and 75% of the pulmonary volume (FEF25-75%) at 3 months.
FEF25-75% at 6 months | 6 months
  Pulmonary function will be measured by forced expiratory flow at 25 and 75% of the pulmonary volume (FEF25-75%) at six months.
FEV1/FVC ratio at baseline | baseline
  FEV1/FVC ratio will be calculated at baseline. The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second (FEV1) to the forced vital capacity (FVC) of the lungs.
FEV1/FVC ratio at 3 months | 3 months
  FEV1/FVC ratio will be calculated at 3 months. The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second (FEV1) to the forced vital capacity (FVC) of the lungs.
FEV1/FVC ratio at 6 months | 6 months
  FEV1/FVC ratio will be calculated at 6 months. The FEV1/FVC ratio is the ratio of the forced expiratory volume in the first one second (FEV1) to the forced vital capacity (FVC) of the lungs.
FOT at baseline. | baseline
  Forced Oscillation Technique (FOT) will be measured at baseline. Forced Oscillation Technique (FOT) measures lung impedance during tidal breathing.
FOT at 3 months. | 3 months
  Forced Oscillation Technique (FOT) will be measured at 3 months. Forced Oscillation Technique (FOT) measures lung impedance during tidal breathing.
FOT at 6 months. | 6 months
  Forced Oscillation Technique (FOT) will be measured at 6 months. Forced Oscillation Technique (FOT) measures lung impedance during tidal breathing.

SECONDARY OUTCOMES:
FACIT score at baseline and monthly on therapy | 6 months
  assess the effect of increasing the dose of IGRT on the patients' well-being by quantitating their fatigue level. Scores range from zero (no fatigue) to 52 (maximum fatigue/worse outcome).
PADQOL-16 at baseline and monthly on therapy | 6 months
  assess the effect of increasing the dose of IGRT on the patients' well-being by quantitating their quality of life. Scores range from zero (no impairment) to 32 (maximum impairment/worse outcome).
St. George's Respiratory Questionnaire at baseline and monthly on therapy | 6 months
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from zero (no impairment) to 100 (maximum impairment/worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Harry Schroeder, MD/PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Community Health 20, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No